CLINICAL TRIAL: NCT04804371
Title: Combined 68Ga-DOTATATE and 18F-FDG PET/CT Imaging in Patients With Well-differentiated, G2-G3, Gastroenteropancreatic (GEP)-Neuroendocrine Tumors (NETs) - A Pilot Study
Brief Title: Dual Tracer (68Ga-DOTATATE and 18F-FDG) PET Imaging in G2 & G3 Gastroenteropancreatic Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Neuroendocrine Tumour Society (CNETS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-5920
Record Dates: First submitted 2021-03-03; First posted 2021-03-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: Histologically proven well diff GEP NET, G2-3, Ki 67 ≥3% (or mitotic index ≥2 mitosis/10HPF).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FDG PETCT scan (Other): 18F-FDG tracer (5 MBq/kg body weight of FDG; up to 550 MBq) will be injected into the intravenous
  Interventions: Drug: F18-FDG

INTERVENTIONS:
Drug: F18-FDG — Evaluate FDG uptake

SUMMARY:
The variable clinical outcome of patients with G2 & G3 well diff GEP-NETs makes the selection of an optimal treatment strategy challenging.

Initial data suggests that high DOTATATE uptake and low FDG uptake are suggestive of low grade disease, with an indolent course.

Conversely, low DT uptake and high FDG uptake are suggestive of high-grade/ aggressive disease.

G2/3 GEP NETs may be biologically diverse; clinically relevant cohort for dual-tracer PET imaging.

Our secondary objectives are

1. To determine the distribution of PETNET scores derived from 18F-FDG & 68Ga-DT PET in patients with G2 & G3 well diff GEP-NETs.
2. To determine the proportion of patients in whom the addition of 18F-FDG PET data results in a change in planned clinical management.

To assess intra-individual variability in SSTR expression & glucose metabolism (as seen on DT and FDG PET) across different tumor sites within the same patient.

2) To determine whether a correlation exists between tumor texture features on 68Ga-DT & FDG PET to tumor grade and Ki 67 index.

3) To assess for an association between tumor texture features on 68Ga-DT PET and glucose metabolism; and/or an association between tumor texture features on FDG PET and SSTR expression.

DETAILED DESCRIPTION:
The variable clinical outcome of patients with G2 and G3 well differentiated GEP-NETs makes the selection of an optimal treatment strategy challenging.

A subject with 68Ga-DOTATATE uptake on all lesions without FDG uptake is likely to have low-grade, metabolically inactive disease, leading to an indolent disease course and may also be a predictive biomarker in subjects being considered for PRRT.

Conversely, avidity on 18F-FDG PET/CT and non-avidity on 68Ga-DOTATATE may indicate a high-grade NET, and would predict resistance to PRRT, suggesting that a more "aggressive" approach with systemic chemotherapy might be beneficial.

Therefore, the prospective assessment of PETNET score in patients with G2 or G3 GEP NETs, which may be biologically diverse is the most clinically relevant group for dual-tracer PET imaging.

Primary Objectives:

1. To determine the distribution of PETNET scores derived from 18F-FDG and 68Ga-DOTATATE PET/CT in patients with G2 and G3 well differentiated GEP-NETs.
2. To determine the proportion of patients in whom the addition of 18F-FDG PET/CT data results in a change in planned clinical management.

Secondary Objectives:

1. mTo determine whether there is intra-individual variability in somatostatin receptor expression and glucose metabolism (as seen on DOTATATE PET and FDG PET, respectively) across different tumor sites within the same patient.
2. To determine whether a correlation exists between tumor texture features on 68Ga-DOTATATE PET and FDG PET to tumor grade and Ki67 index.
3. To assess if an association exists between tumor texture features on 68Ga-DOTATATE PET and glucose metabolism; and/or an association between tumor texture features on FDG PET and somatostatin receptor expression.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent prior to any study-related procedures,
2. Is a male or a female of 18 years of age or older.
3. Patients who already had/scheduled for a 68Ga-DOTATATE PET/CT scan.
4. Has a gastro entero-pancreatic neuroendocrine neoplasm confirmed by histological criteria. Patients with unknown primaries clinically thought to be from gastroenteropancreatic source shall be eligible.
5. Has a well differentiated tumour Grade 2-3 (WHO 2017).
6. Has a tumour with a proliferation index (Ki67 ≥3%) or in samples where the Ki67 antigen cannot be reliably quantified, a mitotic index ≥2 mitosis/10HPF (high power fields)
7. Treatment naïve patients and/or patient who have received any number of prior systemic therapy lines for metastatic disease and/or locally advanced inoperable tumor.
8. Willing and able to comply with all study requirements, including timing and/or nature of required assessments.
9. Women of child-bearing age will undergo a urine test to exclude pregnancy prior to PET.

Exclusion Criteria:

1. Patients with known lung neuroendocrine tumours or other proven non gastroenteropancreatic histologies are not eligible.
2. Patients with any known hypersensitivity to FDG.
3. Has a well differentiated neuroendocrine tumour Grade 1 (WHO 2017).
4. Has a poorly differentiated neuroendocrine carcinoma (WHO 2017).
5. Mixed neuroendocrine and non-neuroendocrine cancer
6. Has any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
7. Any patient who is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Discordance in tracer uptake: | 2 years
  Discordance in tracer uptake as assessed by PETNET score distribution: Proportion of patients with PETNET score of P1/P2 (no or low FDG uptake) vs those with P3-P5 (moderate or high FDG uptake).
Impact to patient management: | 2 years
  Impact of the addition of FDG PET to patient management as assessed by rate of clinical management changed after the addition of 18F-FDG PET/CT to 68Ga-DOTATATE PET/CT.

SECONDARY OUTCOMES:
Intraindividual tumor heterogeneity: | 2 years
  Assessment of tumor heterogeneity by measuring the proportion of patients with variable PET NET score at different tumor sites (intraindividual variability).
Tumor texture geatures as predictors of tumor grade: | 2 years
  To determine whether tumor texture features on PET correlate with tumor grade and/or Ki-67 index.
Tumor texture features as predictors of tumor metabolism and somatostatin receptor expression: | 2 years
  To determine whether tumor texture features on 68Ga-DOTATATE PET correlate with glucose metabolism (as measured semiquantitatively with SUV on FDG PET); and/or whether tumor texture features on FDG PET correlate with somatostatin receptor expression (as measured semiquantitatively with SUV on 68Ga-DOTATATE PET).

CONTACTS AND LOCATIONS:
Overall Officials: Ur Metser, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada